CLINICAL TRIAL: NCT04033939
Title: A Phase I, Placebo and Positive-controlled, Dose-escalation Study to Determine the Safety, Pharmacodynamics and Pharmacokinetics of a Single Intravenous Injection of HSK3486 in Healthy Subjects
Brief Title: A Study Evaluating the Safety, Pharmacodynamics and Pharmacokinetics of HSK3486 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486Australia-01
Record Dates: First submitted 2019-07-04; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Masking Description: Following Screening, subjects who meet the inclusion/exclusion criteria will be assigned a subject number in the order in which they are enrolled in the study. The subject number will determine the allocation of treatment as per the randomization list which will be generated by INCResearch Australia Pty Ltd and provided to the pharmacist. Cohorts 1 and 2 are a placebo controlled design, with open-labelling for the sentinel subjects and double-blind thereafter. Cohorts 3 to 8 are an open-label, positive controlled design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK3486-01 (Experimental): Randomized to receive HSK3486 (0.016mg/kg,0.064mg/kg )as a single IV injection. HSK3486-01 was blinded.(2 HSK3486-01: 1 Placebo-01)
  Interventions: Drug: HSK3486
- Placebo-01 (Placebo Comparator): Randomized to receive placebo (0.016mg/kg,0.064mg/kg )as a single IV injection. placebo-01 was blinded.(2 HSK3486-01: 1 Placebo-01)
  Interventions: Drug: Placebo
- HSK3486-02 (Experimental): Randomized to receive either HSK3486（0.128mg/kg,0.192mg/kg,0.288mg/kg,0.432mg/kg,0.540mg/kg,0.648mg/kg,0.810mg/kg) as a single IV injection. HSK3486-02 was open-label.(5 HSK3486-02: 1 propofol-02)
  Interventions: Drug: HSK3486
- Propofol-02 (Active Comparator): Randomized to receive propofol (2.5mg/kg) as a single IV injection. Propofol-02 was open-label.(5 HSK3486-02: 1 propofol-02)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486
  Arms: HSK3486-01; HSK3486-02
Drug: Propofol
  Arms: Propofol-02
Drug: Placebo
  Arms: Placebo-01

SUMMARY:
This is the first clinical trial of HSK3486 and will be conducted in healthy volunteers to determine the safety, tolerability (including pain on injection), and PK(only to be assessed for subjects who are randomized to HSK3486 in Cohorts 3 to 8)and PD and profiles of HSK3486 administered as a single IV injection.

Results from this study will supports further clinical development of HSK3486. This study will be performed in compliance with the protocol, International Conference on Harmonization Good Clinical Practice (ICH GCP) and local regulatory requirements. Aspects of the study concerned with the investigational product will meet the requirements of Good Manufacturing Practice (GMP).

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 - 49 years (inclusive).
* In general good health without clinically significant (CS) medical history.
* American Society of Anesthesiologists (ASA) Physical Status Classification of I or II.
* Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive).
* Negative screen for drugs of abuse, alcohol, Hepatitis B surface antigen (HBs-Ag), Hepatitis C Virus antibody (HCV-Ab) and Human Immunodeficiency Virus (HIV) at screening; and drugs of abuse, alcohol pre dose on Day -1.
* Normal or non-clinically significant (NCS) findings on a physical examination, 12-lead electrocardiogram (ECG) and vital signs (respiration rate between 12 and 20 breaths per minute, blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats per minute, temperature between 35.8°C and 37.5°C and pulse oximetry values > 95% on room air).
* Clinical laboratory values within the normal limits as defined by the clinical laboratory samples, unless the Principal Investigator (PI) decided that out-of-range values were not CS.
* Able to provide written informed consent.
* Willing and able to follow study instructions and likely to complete all study requirements.
* Suitable venous and arterial access.

Exclusion Criteria:

* History of allergy or sensitivity to: propofol, components of Fresofol 1% MCT/LCT propofol, or HSK3486 (excipients soy bean oil, glycerine, triglycerides, purified egg phospholipids, sodium oleate and sodium hydroxide), or plain lignocaine.
* History of CS problems with general anesthesia.
* Current smoker, or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within 2 months prior to screening.
* History of excessive alcohol intake (more than four standard drinks daily, on average) or use of recreational drugs within the last 3 months.
* Use of prescription or over the counter medications within 7 days of Investigational Product administration, with the exception of simple analgesics such as paracetamol and oral non-steroidal antiinflammatory agents.
* Standard donation of blood within 30 days of the study.
* Donation of plasma or participation in a plasmapheresis program within 7 days preceding this study.
* Receipt of any investigational study drug within 30 days prior to screening.
* Unable to fast for the 6 hours prior to Investigational Product administration.
* Clinically significant (as judged by the Investigator) presence of acute illness (e.g. gastrointestinal illness, infection such as influenza, upper respiratory tract infection) at admission to the clinical study unit.
* Anticipated need for surgery or hospitalization during the study.
* Anatomical abnormality that would potentially interfere with airway management under unconscious sedation or anesthesia.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04-13 (Actual); Primary Completion 2014-11-11 (Actual); Study Completion 2015-05-04 (Actual)

PRIMARY OUTCOMES:
Safety by measurement of Adverse Events | First dose of study drug on day 1

SECONDARY OUTCOMES:
Median effective dose (ED50) | From first dose of study drug until fully alert on day 1
Peak concentration (Cmax) | From the start of administration to 48 hours after administration
Time to plasma peak concentration(Tmax) | From the start of administration to 48 hours after administration
Terminal elimination half life (t1/2z) and mean residence time (MRT) | From the start of administration to 48 hours after administration
Mean residence time (MRT) | From the start of administration to 48 hours after administration
Area Under the Curve (AUC0-30min, AUC0-1h, AUC0-last, and AUC0-inf) | From the start of administration to 48 hours after administration
Total clearance (CL) | From the start of administration to 48 hours after administration